CLINICAL TRIAL: NCT02078934
Title: Endoscopic Gastric Plication for Weight Loss in Morbidly Obese Patients Prior to Incisional Hernia
Brief Title: Endoscopic Gastric Plication for Weight Loss in Morbidly Obese Patients Prior to Incisional Hernia Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding for recruitment.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endoscopic Gastric Plication
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Morbid Obesity; Weight Loss; Complex Incisional Hernias
Keywords: Surgical Endoscopy; Morbid Obesity; Weight Loss; Bariatrics; Complex incisional hernia with mesh
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight Loss (Experimental): Patients with complex incisional/ventral hernias who are too obese to undergo hernia repair.
  Interventions: Procedure: Endoscopic Gastric Plication

INTERVENTIONS:
Procedure: Endoscopic Gastric Plication — Evaluate the efficacy of endoscopic suturing for weight loss
  Other Names: Endoscopic Sleeve Plication; Apollo Suturing

SUMMARY:
Incisional hernias occur in nearly 20% of all laparotomy incisions accounting for almost 400,000 ventral hernia repairs annually in the United States. There is an even higher incidence of incisional hernia recurrence after prior repair if the patient is obese. Each subsequent hernia repair leads to increased morbidity and durability. It is not infrequent that many surgeons will advise overweight or obese patients to lose substantial weight prior to complex incisional hernia repair.

However, it is quite difficult for any individual to lose more than 8 pounds a month in a safe, rapid, and sustainable fashion. This is based on losing 2 lbs. per week utilizing diet and exercise alone. Many patients with incisional hernia are physically debilitated that they cannot engage in any substantial physical activity to lose weight. Traditional laparoscopic bariatric surgery (i.e. Roux-en-Y gastric bypass (RYGB) and SG), while feasible, is a technically challenging endeavor since prior abdominal surgeries increase the amount of intra-abdominal adhesions. Furthermore, there is still a subset of patients who are not candidates for laparoscopic weight loss surgery because of inability to tolerate pneumoperitoneum due to underlying physiologic dysfunction.

- Novel minimally invasive endoscopic technique may help obese patients with an incisional hernia lose weight in a safe and rapid fashion. Early case reports and small case series on gastric bypass revision utilizing such endoscopic technique have shown promise in efficacious weight loss. There have been reports of achieving nearly 20-25% excess weight loss.

Abu Dayyeh and colleagues have also demonstrated that endoscopic gastric plication as a primary weight loss procedure is feasible, but their reported follow-up was only 3 months.8 Brethauer, et al. from Cleveland Clinic performed transoral gastric volume reduction for weight management in 18 patients (TRIM TRIAL). They utilized the Restore Suturing System (Restore device) and reported a mean decrease in BMI of -4.0 ± 3.5 kg/m2. Mean excess weight loss was 27.7% ± 21.9% with no reports of adverse events.9 There have also been reports of not only weight loss but improved insulin sensitivity and secretion.10 Laparoscopic gastric greater curvature plication afforded a mean 50.7% excess weight loss at 12 months.11

The intent of this study is not to demonstrate endoscopic suturing to be a primary option for weight-loss surgery. Preliminary reports have shown such procedure is technically feasible but not durable and the effects of the procedure varied widely among the study participants.12 The investigators view this technology as a bridge for morbidly obese patients, who will need subsequent surgery for another surgical disease, to improve their body habitus and decrease their postoperative morbidity and mortality. The aims of the investigators study are:

* Feasibility of endoscopic gastric sleeve plication
* Define the technical aspects of endoscopic suturing for sleeve plication
* Provide long-term follow-up for both weight loss and resolution of their co-morbidities
* Time from the endoscopic procedure to their incisional hernia repair
* Photographic evidence of the stomach after endoscopic plication during the incisional hernia repair

There are several advantages for the proposed study. First it avoids entering the intra-abdominal cavity. Second, the procedure is performed solely with sutures obviating the need for stapling which may increase the risk of gastric leak from the staple line.13 Lastly, it avoids placing endoscopic intra-luminal devices such as intragastric balloons or duodenal-jejunal sleeves. Limiting factor of such devices is a high rate of premature device withdrawal due to intolerance. Furthermore, their effects are short-lived as most devices will need to be removed by 12 weeks and they only offer a mean 23.6% excess weight loss.13, 14

The implications of this study can be far-reaching. Once efficacy is demonstrated where enough weight loss is achieved that patients can safely and quickly undergo their incisional hernia surgery, the investigators can then conduct a retrospective case-control cross-matched study to further delineate its true benefit. If there is a true benefit, then a randomized control study can be employed in the future.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ³35 kg/m2
* Documented incisional hernia
* Age ≥ 18 years old

Exclusion Criteria:

* Prior gastric surgery
* Prior bariatric surgery
* Gastroesophageal reflux disease (GERD)
* Enterocutaneous fistula (ECF)
* Unable to tolerate general anesthesia
* Portal Hypertension
* Underlying coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 1 Year
  We will track patient's weight loss after their endoscopic bariatric surgery.

SECONDARY OUTCOMES:
Time to Hernia Repair | 1 year
  See the time it takes for the patient from the endoscopic surgery to the actual hernia surgery.

OTHER OUTCOMES:
Hernia Repair | 3 years
  Success of hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J. Rogers, MD, Principal Investigator — University of California, San Francisco; Jonathan T Carter, MD, Principal Investigator — University of California, San Francisco; Matthew YC Lin, MD, Principal Investigator — University of California, San Francisco; John P Cello, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Le Huu Nho R, Mege D, Ouaissi M, Sielezneff I, Sastre B. Incidence and prevention of ventral incisional hernia. J Visc Surg. 2012 Oct;149(5 Suppl):e3-14. doi: 10.1016/j.jviscsurg.2012.05.004. Epub 2012 Nov 9. PMID 23142402
- [Background] Funk LM, Perry KA, Narula VK, Mikami DJ, Melvin WS. Current national practice patterns for inpatient management of ventral abdominal wall hernia in the United States. Surg Endosc. 2013 Nov;27(11):4104-12. doi: 10.1007/s00464-013-3075-4. Epub 2013 Jul 17. PMID 23860608
- [Background] Cote GA, Edmundowicz SA. Emerging technology: endoluminal treatment of obesity. Gastrointest Endosc. 2009 Nov;70(5):991-9. doi: 10.1016/j.gie.2009.09.016. PMID 19879407
- [Background] Familiari P, Costamagna G, Blero D, Le Moine O, Perri V, Boskoski I, Coppens E, Barea M, Iaconelli A, Mingrone G, Moreno C, Deviere J. Transoral gastroplasty for morbid obesity: a multicenter trial with a 1-year outcome. Gastrointest Endosc. 2011 Dec;74(6):1248-58. doi: 10.1016/j.gie.2011.08.046. PMID 22136774
- [Background] Brethauer SA, Chand B, Schauer PR, Thompson CC. Transoral gastric volume reduction as intervention for weight management: 12-month follow-up of TRIM trial. Surg Obes Relat Dis. 2012 May-Jun;8(3):296-303. doi: 10.1016/j.soard.2011.10.016. Epub 2011 Nov 9. PMID 22178565
- [Background] Brethauer SA, Chand B, Schauer PR, Thompson CC. Transoral gastric volume reduction for weight management: technique and feasibility in 18 patients. Surg Obes Relat Dis. 2010 Nov-Dec;6(6):689-94. doi: 10.1016/j.soard.2010.07.012. Epub 2010 Aug 6. PMID 20947451
- [Background] Abu Dayyeh BK, Rajan E, Gostout CJ. Endoscopic sleeve gastroplasty: a potential endoscopic alternative to surgical sleeve gastrectomy for treatment of obesity. Gastrointest Endosc. 2013 Sep;78(3):530-5. doi: 10.1016/j.gie.2013.04.197. Epub 2013 May 24. PMID 23711556